CLINICAL TRIAL: NCT01523782
Title: An Escalating Dose Phase IIa Study of L-Asparaginase Encapsulated in Erythrocytes (GRASPA®) in Association With Polychemotherapy During Induction Phase for Treatment of Elderly Patients With Acute Lymphoblastic Leukaemia (ALL), Aged 55 Years and Over, With Philadelphia Chromosome-negative (ALL Ph-)
Brief Title: Administration of GRASPA (Suspension of Erythrocytes Encapsulating L-asparaginase) in Elderly Patients With First Line Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ERYtech Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GRASPALL/GRAALLSA2-2008
Record Dates: First submitted 2012-01-16; First posted 2012-02-01 (Estimated); Results first posted 2018-06-14 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2018-06

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Acute Lymphoblastic leukemia; Elderly patient; Asparaginase
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- GRASPA 50 IU/kg (Experimental): Each patient will receive GRASPA 50 IU/kg at day 3 of the induction 1 phase. If no toxicity related to investigational product is observed and if the patient's state of health allows it, a second injection, at the identical dose, will be administered at Day 6 of Induction 2 phase.
  Interventions: Drug: GRASPA
- GRASPA 100 IU/kg (Experimental): Each patient will receive GRASPA 100 IU/kg at day 3 of the induction 1 phase. If no toxicity related to investigational product is observed and if the patient's state of health allows it, a second injection, at the identical dose, will be administered at Day 6 of Induction 2 phase
  Interventions: Drug: GRASPA
- GRASPA 150 IU/kg (Experimental): Each patient will receive GRASPA 150 IU/kg at day 3 of the induction 1 phase. If no toxicity related to investigational product is observed and if the patient's state of health allows it, a second injection, at the identical dose, will be administered at Day 6 of Induction 2 phase
  Interventions: Drug: GRASPA

INTERVENTIONS:
Drug: GRASPA — Each patient will receive GRASPA at day 3 of the induction 1 phase. If no toxicity related to investigational product is observed and if the patient's state of health allows it, a second injection, at the identical dose, will be administered at Day 6 of Induction 2 phase

SUMMARY:
The main purpose of this study is to determine the maximum tolerated and efficient dose of GRASPA® in combination with polychemotherapy treatment of elderly patients with ALL, 55 years and over, Philadelphia chromosome-negative (ALL Ph-).

DETAILED DESCRIPTION:
This open label, non randomised, multicentric and national phase IIa study was designed to evaluate the safety and efficacy of GRASPA®, a suspension of red blood cells encapsulating E. Coli L-asparaginase, at different doses and in combination with the polychemotherapy regimen recommended by the European Working Group on Adult ALL (EWALL) for frontline therapy of patients with ALL Ph-, aged 55 years old and over. Patients with a good performance status (WHO score ≤2) and a newly diagnosed ALL Ph- were treated with the backbone polychemotherapy consisting of a first 4-week induction phase comprising dexamethasone, vincristine and idarubicin, a second 4-week induction phase including cyclophosphamide, cytarabine, a 6-month consolidation phase consisting of 6 alternating cycles with methotrexate, asparaginase and folinic acid (cycles 1, 3 and 5) and high-dose cytarabine (cycles 2, 4 and 6) with Granulocyte colony stimulating factor (G-CSF) support followed by a 16-month maintenance period with mercaptopurine, methotrexate and vincristine/dexamethasone pulses. GRASPA® was administered on day 3 of induction 1 and on day 6 of induction 2 of the chemotherapy regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥55 years old
* With newly diagnosed ALL without prior treatment
* Capable to receive polychemotherapy (World Health Organization (WHO) performance status ≤2)
* With or without meningeal disease
* Having signed an Informed Consent Form
* Subscribed to social security insurance

Exclusion Criteria:

* ALL translocation(9;22) and/or BCR-ABL (Breakpoint Cluster Region-Abelson) positive
* Performance status incompatible with chemotherapy treatment (WHO score >2)
* Patient presenting with a general or visceral contraindication to intensive treatment including :

  * Cardiac insufficiency defined as Left Ventricular Ejection Fraction <50% of the theoretical value
  * Plasma creatinine concentration 2 times greater than the upper limit of laboratory ranges, except if related to ALL
  * Aspartate aminotransferase (ASAT) or alanine aminotransferase (ALAT) levels 5 times greater than the upper limit of laboratory ranges, except if related to ALL
  * Patient with another evolutive cancer other than ALL
  * Severe evolutive infection, or Human Immunodeficiency Virus (HIV) seropositive or, active hepatitis related to B or C viral infection
* Prior treatment with L-asparaginase (irrespective of the form)
* History of grade 3 transfusional incident (life threatening)
* Patient presenting rare and/or dangerous anti-erythrocyte antibodies thus leading to the unavailability of phenotype compatible Red Blood Cells Concentrate
* Patient included in another clinical trial during the last 4 weeks

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-04; Primary Completion 2011-01 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde Hunault-Berger, Professor, Principal Investigator — University Hospital, Angers

IPD SHARING:
Plan to Share IPD: No
Not applicable for this study

REFERENCES:
- [Derived] Hunault-Berger M, Leguay T, Huguet F, Lepretre S, Deconinck E, Ojeda-Uribe M, Bonmati C, Escoffre-Barbe M, Bories P, Himberlin C, Chevallier P, Rousselot P, Reman O, Boulland ML, Lissandre S, Turlure P, Bouscary D, Sanhes L, Legrand O, Lafage-Pochitaloff M, Bene MC, Liens D, Godfrin Y, Ifrah N, Dombret H; Group for Research on Adult Acute Lymphoblastic Leukemia (GRAALL). A Phase 2 study of L-asparaginase encapsulated in erythrocytes in elderly patients with Philadelphia chromosome negative acute lymphoblastic leukemia: The GRASPALL/GRAALL-SA2-2008 study. Am J Hematol. 2015 Sep;90(9):811-8. doi: 10.1002/ajh.24093. PMID 26094614

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GRASPA 50 IU/kg | GRASPA 100 IU/kg | GRASPA 150 IU/kg
Started | 3 | 13 | 14
Completed | 2 | 13 | 9
Not Completed | 1 | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GRASPA 50 IU/kg | GRASPA 100 IU/kg | GRASPA 150 IU/kg | Total
Number analyzed (Participants) | 3 | 13 | 14 | 30
Age, Continuous [Mean (Full Range); unit: years] | 68.33 [65.0 to 72.0] | 66.92 [59.0 to 77.0] | 67.00 [61.0 to 77.0] | 67.10 [59.0 to 77.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 8 | 16
  Male | 1 | 7 | 6 | 14
Region of Enrollment [Number; unit: participants]
  France | 3 | 13 | 14 | 30

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Primary Endpoint - Percentage of Patients Responding to Treatment
Description: The main evaluation criterion is a composite efficacy/toxicity criterion. Efficacy, assessed during induction 1: percentage of patients responding to treatment, i.e. with plasma Asn concentration ≤2µM (depleted), for a duration of at least 7 days after the administration of GRASPA®
Time Frame: 7 days after the first administration of GRASPA® during Induction 1
Measure: Count of Participants; unit: Participants
Arm/Group | GRASPA 50 IU/kg | GRASPA 100 IU/kg | GRASPA 150 IU/kg
Number analyzed (Participants) | 3 | 13 | 14
Participants | 0 | 11 | 10

2. Primary Outcome: Safety Endpoint - DLTs Assessed During Induction 1 and Induction 2
Description: Safety: Toxicity, assessed during Induction 1 and Induction 2: according to NCI-CTCAE v3.0 August 2006, with Dose Limiting Toxicities (DLT) defined as: Grade 2 to 4 pancreatic toxicity, Grade 3 or 4 hepatic toxicity, allergic toxicity or deep cerebral thrombosis, known as potentially related to L-asparaginase; hematological toxicity defined as bone marrow blast free aplasia, 30 days following the last injection of chemotherapy, all other Grade 4 toxicities.
Time Frame: Induction 1 and Induction 2
Measure: Number; unit: DLTs
Arm/Group | GRASPA 50 IU/kg | GRASPA 100 IU/kg | GRASPA 150 IU/kg
Number analyzed (Participants) | 3 | 13 | 14
DLTs | 0 | 5 | 17

3. Secondary Outcome: Plasma Concentrations of Asparagine
Description: Mean plasma concentration of asparagine over time. Participants who were Below the Lower Limit of Quantification (BLLQ) were assigned a value of 0.51 μmol/L.
Time Frame: Induction 1 & Induction 2
Population: The participant numbers in some of the rows below differ from the overall participant numbers analyzed because we are missing the values from some of those time points.
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | GRASPA 50 IU/kg | GRASPA 100 IU/kg | GRASPA 150 IU/kg
Number analyzed (Participants) | 3 | 13 | 14
μmol/L
  Induction 1, Day 3 | 60.86 (9.38) | 46.74 (21.44) | 42.33 (10.98)
  Induction 1, Day 4 | 0.51 (0) | 0.51 (0) | 0.51 (0)
  Induction 1, Day 10 | 17.48 (11.46) | 1.78 (3.39) | 3.11 (4.05)
  Induction 1, Day 17: number analyzed (Participants) | 3 | 13 | 13
  Induction 1, Day 17 | 16.33 (9.62) | 10.05 (8.10) | 9.30 (7.39)
  Induction 1, Day 22-28: number analyzed (Participants) | 2 | 11 | 12
  Induction 1, Day 22-28 | 24.55 (1.60) | 20.35 (10.60) | 18.76 (8.74)
  Induction 2, Day 6: number analyzed (Participants) | 2 | 12 | 9
  Induction 2, Day 6 | 45.39 (1.24) | 28.11 (9.74) | 27.16 (14.45)
  Induction 2, Day 7: number analyzed (Participants) | 2 | 12 | 9
  Induction 2, Day 7 | 9.41 (12.59) | 9.44 (16.23) | 0.51 (0)
  Induction 2, Day 13: number analyzed (Participants) | 2 | 11 | 9
  Induction 2, Day 13 | 29.47 (34.69) | 10.37 (11.16) | 3.79 (6.58)
  Induction 2, Day 20: number analyzed (Participants) | 2 | 11 | 9
  Induction 2, Day 20 | 34.20 (8.48) | 13.71 (10.40) | 12.91 (8.17)
  Induction 2, Day 22 to D28: number analyzed (Participants) | 2 | 10 | 8
  Induction 2, Day 22 to D28 | 46.22 (28.92) | 17.27 (12.12) | 17.23 (4.77)

4. Secondary Outcome: Plasma Concentrations of Aspartic Acid
Description: Mean plasma concentration of aspartic acid over time.
Time Frame: Induction 1 and Induction 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | GRASPA 50 IU/kg | GRASPA 100 IU/kg | GRASPA 150 IU/kg
Number analyzed (Participants) | 3 | 13 | 14
μmol/L
  Induction 1, D3 | 1.91 (0.28) | 2.38 (4.39) | 3.59 (5.03)
  Induction 1, D4 | 11.08 (4.14) | 5.22 (1.81) | 8.11 (5.50)
  Induction 1, D10 | 17.93 (3.65) | 16.47 (6.17) | 13.51 (5.16)
  Induction 1, D17: number analyzed (Participants) | 3 | 13 | 13
  Induction 1, D17 | 3.76 (1.39) | 10.60 (6.02) | 8.43 (4.58)
  Induction 1, D22-28: number analyzed (Participants) | 2 | 12 | 13
  Induction 1, D22-28 | 5.17 (1.82) | 10.27 (9.88) | 6.93 (5.31)
  Induction 2, D6: number analyzed (Participants) | 2 | 12 | 9
  Induction 2, D6 | 2.32 (0.63) | 4.17 (4.31) | 5.08 (3.35)
  Induction 2, D7: number analyzed (Participants) | 2 | 12 | 9
  Induction 2, D7 | 12.06 (6.36) | 6.35 (3.67) | 7.59 (3.45)
  Induction 2, D13: number analyzed (Participants) | 2 | 11 | 9
  Induction 2, D13 | 9.07 (8.92) | 9.82 (6.52) | 10.07 (5.19)
  Induction 2, D20: number analyzed (Participants) | 2 | 11 | 9
  Induction 2, D20 | 2.56 (0.37) | 8.39 (6.58) | 7.06 (5.28)
  Induction 2, D22-28: number analyzed (Participants) | 2 | 10 | 9
  Induction 2, D22-28 | 3.37 (1.00) | 11.04 (8.66) | 6.32 (4.75)

5. Secondary Outcome: Plasma Concentrations of Glutamine
Description: Mean glutamine concentration over time.
Time Frame: Induction 1 and Induction 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | GRASPA 50 IU/kg | GRASPA 100 IU/kg | GRASPA 150 IU/kg
Number analyzed (Participants) | 3 | 13 | 14
μmol/L
  Induction 1, D3 | 558.78 (158.02) | 484.19 (137.05) | 432.07 (69.93)
  Induction 1, D4 | 616.13 (184.59) | 494.76 (142.95) | 463.03 (117.79)
  Induction 1, D10 | 576.86 (172.51) | 521.86 (180.41) | 447.07 (159.93)
  Induction 1, D17: number analyzed (Participants) | 3 | 13 | 13
  Induction 1, D17 | 384.12 (28.05) | 344.03 (102.95) | 266.08 (71.48)
  Induction 1, D22-28: number analyzed (Participants) | 2 | 12 | 13
  Induction 1, D22-28 | 394.53 (21.50) | 422.76 (175.67) | 393.87 (78.01)
  Induction 2, D6: number analyzed (Participants) | 2 | 12 | 9
  Induction 2, D6 | 508.99 (17.53) | 436.71 (140.02) | 426.28 (72.15)
  Induction 2, D7: number analyzed (Participants) | 2 | 12 | 9
  Induction 2, D7 | 553.63 (71.15) | 498.41 (131.33) | 445.00 (145.95)
  Induction 2, D13: number analyzed (Participants) | 2 | 11 | 9
  Induction 2, D13 | 517.42 (50.94) | 467.52 (136.17) | 456.52 (113.75)
  Induction 2, D20: number analyzed (Participants) | 2 | 11 | 9
  Induction 2, D20 | 436.17 (15.72) | 406.62 (101.32) | 394.51 (69.15)
  Induction 2, D22-28: number analyzed (Participants) | 2 | 10 | 9
  Induction 2, D22-28 | 530.40 (167.13) | 504.97 (117.83) | 441.50 (60.63)

6. Secondary Outcome: Plasma Concentrations of Glutamic Acid.
Description: Mean glutamic acid concentration over time.
Time Frame: Induction 1 and Induction 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | GRASPA 50 IU/kg | GRASPA 100 IU/kg | GRASPA 150 IU/kg
Number analyzed (Participants) | 3 | 13 | 14
μmol/L
  Induction 1, D3 | 49.96 (17.23) | 28.68 (18.01) | 39.87 (49.71)
  Induction 1, D4 | 94.73 (35.53) | 54.38 (29.68) | 52.17 (29.01)
  Induction 1, D10 | 53.58 (6.94) | 31.87 (17.41) | 31.82 (23.20)
  Induction 1, D17: number analyzed (Participants) | 3 | 13 | 13
  Induction 1, D17 | 65.73 (21.31) | 39.71 (27.67) | 31.57 (23.33)
  Induction 1, D22-28: number analyzed (Participants) | 2 | 12 | 13
  Induction 1, D22-28 | 42.83 (2.56) | 46.74 (27.49) | 36.49 (22.90)
  Induction 2, D6: number analyzed (Participants) | 2 | 12 | 9
  Induction 2, D6 | 58.94 (37.41) | 53.88 (29.03) | 55.94 (32.51)
  Induction 2, D7: number analyzed (Participants) | 2 | 12 | 9
  Induction 2, D7 | 77.11 (29.37) | 63.51 (35.37) | 83.98 (49.74)
  Induction 2, D13: number analyzed (Participants) | 2 | 11 | 9
  Induction 2, D13 | 34.70 (9.57) | 53.64 (27.70) | 52.24 (23.91)
  Induction 2, D20: number analyzed (Participants) | 2 | 11 | 9
  Induction 2, D20 | 27.83 (7.63) | 42.86 (20.70) | 35.09 (14.87)
  Induction 2, D22-28: number analyzed (Participants) | 2 | 10 | 9
  Induction 2, D22-28 | 56.21 (1.85) | 47.92 (31.07) | 42.62 (11.94)

7. Secondary Outcome: Cerebral Spinal Fluid Concentrations of Asparagine
Description: Mean cerebral spinal fluid asparagine concentration over time.
Time Frame: Induction 1 and Induction 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | GRASPA 50 IU/kg | GRASPA 100 IU/kg | GRASPA 150 IU/kg
Number analyzed (Participants) | 2 | 12 | 9
μmol/L
  Induction 1, D2: number analyzed (Participants) | 2 | 12 | 8
  Induction 1, D2 | 5.98 (0.63) | 8.35 (3.20) | 6.06 (3.17)
  Induction 1, D9 | 6.57 (2.72) | 1.47 (1.28) | 1.61 (1.09)
  Induction 2, D2: number analyzed (Participants) | 2 | 12 | 6
  Induction 2, D2 | 6.24 (1.07) | 6.42 (2.62) | 7.59 (5.58)
  Induction 2, D9: number analyzed (Participants) | 2 | 11 | 5
  Induction 2, D9 | 5.09 (2.99) | 2.74 (4.24) | 0.52 (0.03)

8. Secondary Outcome: Cerebral Spinal Fluid Concentrations of Aspartic Acid
Description: Mean cerebral spinal fluid aspartic acid concentration
Time Frame: Induction 1 and Induction 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | GRASPA 50 IU/kg | GRASPA 100 IU/kg | GRASPA 150 IU/kg
Number analyzed (Participants) | 2 | 12 | 9
μmol/L
  Induction 1, D2 | .95 (0.00) | .95 (0.00) | .95 (0.01)
  Induction 1, D9 | .95 (0.00) | 1.04 (0.32) | 1.10 (0.46)
  Induction 2, D2: number analyzed (Participants) | 2 | 12 | 6
  Induction 2, D2 | .95 (0.00) | .95 (0.00) | 1.35 (0.98)
  Induction 2, D9: number analyzed (Participants) | 2 | 11 | 5
  Induction 2, D9 | .95 (0.00) | 1.09 (0.26) | .95 (0.00)

9. Secondary Outcome: Cerebral Spinal Fluid Concentrations of Glutamine
Description: Mean cerebral spinal fluid glutamine concentration
Time Frame: Induction 1 and Induction 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | GRASPA 50 IU/kg | GRASPA 100 IU/kg | GRASPA 150 IU/kg
Number analyzed (Participants) | 2 | 12 | 9
μmol/L
  Induction 1, D2 | 270.57 (108.21) | 441.34 (239.50) | 408.56 (116.84)
  Induction 1, D9 | 395.76 (32.50) | 363.40 (142.12) | 360.57 (99.56)
  Induction 2, D2: number analyzed (Participants) | 2 | 12 | 6
  Induction 2, D2 | 345.41 (4.13) | 358.90 (107.03) | 378.14 (70.19)
  Induction 2, D9: number analyzed (Participants) | 2 | 11 | 5
  Induction 2, D9 | 372.56 (15.67) | 420.96 (93.42) | 351.30 (44.86)

10. Secondary Outcome: Cerebral Spinal Fluid Concentrations of Glutamic Acid
Description: Mean cerebral spinal fluid glutamic acid concentration
Time Frame: Induction 1 and Induction 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | GRASPA 50 IU/kg | GRASPA 100 IU/kg | GRASPA 150 IU/kg
Number analyzed (Participants) | 2 | 12 | 9
μmol/L
  Induction 1, D2 | 91.55 (39.44) | 91.98 (85.00) | 61.48 (53.96)
  Induction 1, D9 | 132.53 (15.09) | 71.78 (38.44) | 43.93 (30.53)
  Induction 2, D2: number analyzed (Participants) | 2 | 12 | 6
  Induction 2, D2 | 69.35 (5.70) | 52.89 (24.63) | 41.24 (20.18)
  Induction 2, D9: number analyzed (Participants) | 2 | 11 | 5
  Induction 2, D9 | 62.04 (8.37) | 60.30 (28.32) | 47.02 (39.12)

11. Secondary Outcome: Summary of Free Asparaginase Over Time
Time Frame: Induction 1 and Induction 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | GRASPA 50 IU/kg | GRASPA 100 IU/kg | GRASPA 150 IU/kg
Number analyzed (Participants) | 3 | 13 | 14
U/L
  Induction 1, D3 | 3.33 (0.00) | 3.38 (0.16) | 3.33 (0.00)
  Induction 1, D4 | 2.21 (0.57) | 6.87 (5.77) | 4.96 (2.63)
  Induction 1, D10 | 0.48 (0.09) | 0.53 (0.23) | 0.51 (0.30)
  Induction 1, D17: number analyzed (Participants) | 3 | 13 | 13
  Induction 1, D17 | 0.73 (0.38) | 0.34 (0.10) | 0.42 (0.26)
  Induction 1, D22-28: number analyzed (Participants) | 2 | 13 | 12
  Induction 1, D22-28 | 0.66 (0.11) | 0.59 (0.37) | 0.49 (0.32)
  Induction 2, D6: number analyzed (Participants) | 2 | 12 | 9
  Induction 2, D6 | 3.33 (0.00) | 1.19 (1.03) | 0.52 (0.18)
  Induction 2, D7: number analyzed (Participants) | 2 | 12 | 9
  Induction 2, D7 | 1.47 (1.65) | 3.50 (2.86) | 4.96 (3.78)
  Induction 2, D13: number analyzed (Participants) | 2 | 11 | 9
  Induction 2, D13 | 0.35 (0.02) | 0.52 (0.35) | 0.45 (0.38)
  Induction 2, D20: number analyzed (Participants) | 2 | 11 | 9
  Induction 2, D20 | 0.45 (0.04) | 0.46 (0.42) | 0.24 (0.07)
  Induction 2, D22-28: number analyzed (Participants) | 1 | 10 | 8
  Induction 2, D22-28 | 0.49 (0.00) | 0.68 (0.95) | 0.35 (0.10)

12. Secondary Outcome: Summary of Encapsulated Asparaginase (U/L) Over Time
Time Frame: Induction 1 and Induction 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | GRASPA 50 IU/kg | GRASPA 100 IU/kg | GRASPA 150 IU/kg
Number analyzed (Participants) | 3 | 13 | 14
U/L
  Induction 1, D3 | 72.50 (0.00) | 239.49 (602.11) | 72.50 (0.00)
  Induction 1, D4 | 915.32 (137.09) | 1308.48 (490.99) | 1795.03 (564.74)
  Induction 1, D10 | 579.22 (129.99) | 1105.24 (339.77) | 1309.08 (497.53)
  Induction 1, D17: number analyzed (Participants) | 3 | 13 | 13
  Induction 1, D17 | 402.41 (181.91) | 790.39 (193.78) | 793.97 (291.67)
  Induction 1, D22-28: number analyzed (Participants) | 2 | 13 | 12
  Induction 1, D22-28 | 383.59 (62.77) | 571.49 (225.69) | 629.35 (253.60)
  Induction 2, D6: number analyzed (Participants) | 2 | 12 | 9
  Induction 2, D6 | 72.50 (0.00) | 382.51 (275.00) | 524.37 (164.72)
  Induction 2, D7: number analyzed (Participants) | 2 | 12 | 9
  Induction 2, D7 | 722.57 (120.11) | 1223.20 (323.83) | 1913.32 (788.45)
  Induction 2, D13: number analyzed (Participants) | 2 | 11 | 9
  Induction 2, D13 | 714.90 (49.91) | 1051.64 (285.32) | 1536.06 (401.09)
  Induction 2, D20: number analyzed (Participants) | 2 | 11 | 9
  Induction 2, D20 | 556.00 (52.10) | 745.22 (288.06) | 1191.24 (450.38)
  Induction 2, D22-28: number analyzed (Participants) | 1 | 10 | 8
  Induction 2, D22-28 | 509.20 (0) | 673.64 (307.10) | 813.98 (240.88)

13. Secondary Outcome: Number of Patients Positive for Anti-L-asparaginase Antibodies
Description: Evaluation of the number of patients testing positive for anti-asparaginase antibodies.
Time Frame: Induction 1 and Induction 2
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GRASPA 50 IU/kg | GRASPA 100 IU/kg | GRASPA 150 IU/kg
Number analyzed (Participants) | 3 | 13 | 14
Participants
  Induction 1, D3 | 0 | 0 | 0
  Induction 1, D4 | 0 | 0 | 0
  Induction 1, D22-28: number analyzed (Participants) | 2 | 13 | 12
  Induction 1, D22-28 | 0 | 1 | 1
  Induction 2, D6: number analyzed (Participants) | 0 | 1 | 6
  Induction 2, D6 | 0 | 0 | 1
  Induction 2, D22-28: number analyzed (Participants) | 2 | 11 | 9
  Induction 2, D22-28 | 1 | 4 | 5

14. Secondary Outcome: Number of Participants With Complete Remission (CR) Rate Following Induction 1 and Induction 2
Description: CR was defined using:
  * Clinical criteria: disappearance of clinical signs of acute lymphocytic leukemia (ALL)
  * Blood criteria: neutrophils > 1 G/L and platelets >100 G/L
  * Medullary criteria: normally rich bone marrow and percentage of blasts <5%
Time Frame: 1 and 2 months
Population: 28 patients were analyzed for CR after Induction 1 (2 pts in 50 IU/kg; 13 pts in 100 IU/kg; 13 pts in 150 IU/kg). 22 patients were analyzed for CR after Induction 2 (2 pts in 50 IU/kg; 11 pts in 100 IU/kg; 9 pts in 150 IU/kg).
Measure: Count of Participants; unit: Participants
Arm/Group | GRASPA 50 IU/kg | GRASPA 100 IU/kg | GRASPA 150 IU/kg
Number analyzed (Participants) | 2 | 13 | 13
Participants
  Participants who met CR criteria at Induction 1 | 2 | 10 | 8
  Participants who met CR criteria at Induction 2: number analyzed (Participants) | 2 | 11 | 9
  Participants who met CR criteria at Induction 2 | 2 | 10 | 7

ADVERSE EVENTS:
Time Frame: The period of adverse event (AE) reporting was from the patient inclusion until the end of the product safety follow-up, reached 2 months after the last GRASPA® administration, thus theoretically corresponding to the end of the 2nd cycle of consolidation (Visit V12).
Description: Some Adverse Events were monitored/assessed without regard to the specific Adverse Event Term (i.e. "Gastrointestinal Disorder" and "General Disorder").
Arm/Group | GRASPA 50 IU/kg | GRASPA 100 IU/kg | GRASPA 150 IU/kg
All-Cause Mortality (participants affected / at risk) | 1/3 | 2/13 | 3/14
Serious Adverse Events (participants affected / at risk) | 3/3 | 13/13 | 13/14
Other Adverse Events (participants affected / at risk) | 3/3 | 13/13 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GRASPA 50 IU/kg (N=3) | GRASPA 100 IU/kg (N=13) | GRASPA 150 IU/kg (N=14)
Septic Shock (Infections and infestations) | 0 | 3 | 3
Escherichia sepsis (Infections and infestations) | 1 | 2 | 0
Aspergillosis (Infections and infestations) | 0 | 1 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 1 | 1
Pneumonia herpes viral (Infections and infestations) | 0 | 1 | 0
Leukemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 6 | 5
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 | 3 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 2 | 4
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 | 1 | 0
Antithrombin III decreased (Investigations) | 0 | 0 | 2
Pancreatic enzymes increased (Investigations) | 0 | 0 | 1
Arrythmia (Cardiac disorders) | 1 | 0 | 0
Cytolytic hepatitis (Hepatobiliary disorders) | 0 | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Bacterial Sepsis (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1
Citrobacter infection (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Klebsiella sepsis (Infections and infestations) | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1
Pneumocystitis jroveci infection (Infections and infestations) | 1 | 0 | 0
Pseudomonal sepsis (Infections and infestations) | 0 | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 1
Stenotrophomonas sepsis (Infections and infestations) | 0 | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 2 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cerebrovascualr accident (Vascular disorders) | 0 | 0 | 2
Subarachnoid haemorrhage (Vascular disorders) | 0 | 0 | 1
Subclavian vein thrombosis (Vascular disorders) | 0 | 1 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Faecaloma (Gastrointestinal disorders) | 1 | 0 | 0
Haemmorhoids (Gastrointestinal disorders) | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Generalised oedema (General disorders) | 0 | 0 | 1
Infusion site ulcer (General disorders) | 0 | 1 | 0
Multi-organ failure (General disorders) | 0 | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GRASPA 50 IU/kg (N=3) | GRASPA 100 IU/kg (N=13) | GRASPA 150 IU/kg (N=14)
Antithrombin III decreased (Investigations) | 2 | 7 | 12
Gamma-glutamyltransferase increased (Investigations) | 1 | 6 | 4
Alanine aminotransferase increased (Investigations) | 1 | 4 | 4
Blood glucose increased (Investigations) | 1 | 4 | 4
Blood bilirubin increased (Investigations) | 0 | 6 | 2
Blood fibrinogen decreased (Investigations) | 0 | 3 | 4
Lipase increased (Investigations) | 1 | 2 | 3
Prothrombin level decreased (Investigations) | 0 | 1 | 5
Activated partial thromboplastin time prolonged (Investigations) | 2 | 0 | 3
Blood albumin decreased (Investigations) | 1 | 2 | 1
Pancreatic enzymes increased (Investigations) | 0 | 2 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 1
Septic Shock (Infections and infestations) | 0 | 3 | 3
Aspergillosis (Infections and infestations) | 1 | 2 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 1 | 2
Escherichia sepsis (Infections and infestations) | 1 | 2 | 0
Lung infection (Infections and infestations) | 0 | 1 | 2
Oral herpes (Infections and infestations) | 0 | 2 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1 | 8
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 2 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 4 | 2
Leukemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 6 | 5
Cytolytic hepatitis (Hepatobiliary disorders) | 1 | 3 | 4
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 2 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 2 | 4
Gastrointestinal disorders (Gastrointestinal disorders) | 1 | 3 | 2
Respiratory disorders (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
General disorder (General disorders) | 0 | 3 | 2
Nervous system (Nervous system disorders) | 1 | 2 | 2
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 | 3 | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 2
Vascular disorder (Vascular disorders) | 1 | 2 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less